CLINICAL TRIAL: NCT05738161
Title: A Phase 1, Single Arm Investigator-initiated Study to Investigate the Safety of Combining the Antibody Magrolimab With Standard First Line Platinum-based Chemotherapy (With Cisplatin / Gemcitabine) in Advanced Urothelial Carcinoma
Brief Title: Magrolimab in Combination With Cytotoxic Chemotherapy in Advanced Urothelial Carcinoma
Acronym: MACOCUC-01
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IMP security Issues reported by Sponsor
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-SW-548-6347; 2023-00258 (Other: Swiss Association of Research Ethics Committees)
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Advanced Urothelial Carcinoma
Keywords: Chemotherapy; Antibody Drug Therapy
MeSH Terms: interventions — magrolimab; Cisplatin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Prospective investigator-initiated single-arm, phase 1 clinical trial, risk category C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Magrolimab in combination with Cisplatin and Gemcitabine (Experimental): Magrolimab therapy in combination with standard first line platinum-based chemotherapy (with Cisplatin / Gemcitabine) in advanced urothelial carcinoma.
  Interventions: Drug: Magrolimab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Magrolimab — Magrolimab in combination with cytotoxic chemotherapy in advanced urothelial carcinoma
  Other Names: Hu-5F9-G4
Drug: Cisplatin — Standard first line platinum-based chemotherapy in advanced urothelial carcinoma
  Other Names: L01XA01 Cisplatin
Drug: Gemcitabine — Standard first line platinum-based chemotherapy in advanced urothelial carcinoma
  Other Names: L01BC05 Gemcitabine

SUMMARY:
In their "Magrolimab" research project, the investigators want to find out whether the new drug Magrolimab in combination with conventional chemotherapy is well tolerated and whether survival or progression-free survival improves.

DETAILED DESCRIPTION:
About 10% of the patients with urothelial carcinoma of the bladder present with advanced disease at time of diagnosis. The five-year overall survival is poor (13%) as treatment options are limited to platinum-based chemotherapy and immune checkpoint inhibitors. Therefore, new therapeutic approaches are urgently needed.

Stimulation of the innate immune response to cancer cells using macrophages to attack tumor cells represents a novel approach of cancer immunotherapy. One mechanism used by tumor cells to prevent phagocytosis and thus avoid clearance by the immune system is to up regulate "don't eat me" signals such as CD47. Blockade of CD47 represents a novel immunotherapy allowing the immune system to eliminate cancer cells. Cytotoxic chemotherapy, in particular Gemcitabine, is known to upregulate calreticulin which is a so called "eat me" signal. Consequently, a combination of Gemcitabine with an anit-CD47 antibody could potentiate the tumor-cell killing effects.

Magrolimab is a first-in-class fully humanized monoclonal antibody blocking CD47 and currently investigated as an immunotherapy in solid as well as hematologic malignancies in several phase 1 - 3 clinical trials. Furthermore, Magrolimab as a novel myeloid specific immune checkpoint inhibitor could be the urgently needed new therapeutic weapon for bladder cancer treatment if it proves to add a significant therapeutic benefit to conventional chemotherapy in advanced muscle invasive bladder cancer. The expected benefit of combining chemotherapy with Magrolimab might be manifold:

* It could result in durable systemic anti-cancer responses and subsequently increase disease free and overall survival
* It could increase the response rate and prolong survival in the metastatic setting
* In case of positive results of this trial, the investigators could expand this approach to the peri-operative setting:

  * In the neoadjuvant setting, it could increase the rate of pathologic complete remission (pCR, ypT0) and subsequently reduce the risk of local recurrence and bladder cancer related death
  * In the adjuvant setting, it could induce antitumor immune response in micro metastases and subsequently reduce risk of local recurrence and improve cancer specific survival.

The primary endpoint of the trial is incidence of adverse events (AEs) and laboratory abnormalities according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0 Secondary endpoints are

* PFS from date of dose initiation as determined by investigator assessment per RECIST, Version 1.1
* DOR, defined as time from first documentation of complete response or partial response to the earliest date of documented disease progression, per RECIST, Version 1.1, or death from any cause, whichever occurs first, as determined by investigator assessment
* OS, defined as date of dose initiation to death from any cause.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before trial treatment and prior to any trial specific procedures.
* Male or female age ≥ 18 years.
* Histologically confirmed locally advanced or metastatic predominant urothelial carcinoma of the bladder or the upper urinary tract being considered not suitable for curative multimodality treatment including surgery by a multidisciplinary tumor board. All histological subtypes eligible if urothelial carcinoma predominant (exception: Small cell component).
* ECOG performance status 0-2 within 7 days prior to IMP treatment start.
* Bone marrow function (within 14 days prior to IMP treatment start): Hemoglobin ≥ 100 g/L, absolute neutrophil count ≥ 1.5 x 109/L, platelet count ≥ 100 x 109/L.
* Hepatic function (within 14 days prior to IMP treatment start): Bilirubin ≤ 1.5 x ULN (except for patients with documented history of Gilbert's disease or genetic equivalent ≤ 3.0 x ULN and primarily unconjugated), AST ≤ 2.5 x ULN, ALT ≤ 2.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN.
* Renal function (within 14 days prior to IMP treatment start): eGFR > 60 mL/min/1.73m., according to CKD-EPI formula.
* Cardiac function (within 28 days prior to IMP treatment start): Left Ventricular Ejection Fraction (LVEF) ≥ 50% as determined by echocardiography (ECHO).
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant during trial treatment and 6 months after the last dose of IMP. A negative pregnancy test within 7 days prior to IMP treatment start is required for all women with child-bearing potential.
* Men agree not to father a child during trial treatment and 6 months after the last dose of study drug.
* Measurable disease by CT or MRI as per RECIST 1.1 criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
* Male and female patients of childbearing potential who engage in heterosexual intercourse must agree to use protocol-specified method(s) of contraception.
* Life expectancy at least 12months.
* Willing and able to comply with the requirements and restrictions in this protocol.
* Pre-treatment blood cross-match completed.
* Body weight > 30kg

EXCLUSION CRITERIA:

* Any pathological evidence of small-cell carcinoma component.
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years prior to IMP treatment start, with the exception of adequately treated cervical carcinoma in situ, localized non-melanoma skin cancer or low risk localized prostate cancer (T1-T2a, Gleason <7, PSA <10 ng/ml).
* Concurrent treatment with Prednisone (or equivalent); except for the prophylactic medication before chemotherapy, treatment of acute hypersensitivity reactions, or chronic treatment (initiated > 6 months prior to IMP treatment start) at low dose (≤ 10 mg/day of Prednisone or an equivalent corticosteroid).
* Previous treatment with a PD-1, PD-L1, or CTLA4 inhibitor.
* Previous chemotherapy with Cisplatin and Gemcitabine.
* Treatment with an anticancer biologic agent within 4 weeks prior to IMP treatment start or have had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to IMP treatment start.

(NOTE: Localized non-CNS radiotherapy, previous hormonal therapy with luteinizing hormone releasing hormone [LHRH] agonists for prostate or breast cancer, and treatment with bisphosphonates and Receptor Activator of Nuclear factor KappaB Ligand (RANKL) inhibitors are not criteria for exclusion. There is no required minimum washout period for these therapies. Patients should be recovered from the effects of radiation.)

* Use of other investigational drugs (drugs not marketed for any indication) within 28 days or 5 half-lives (whichever is longer) of IMP treatment start.
* Current participation in another interventional clinical trial. Patients participating in observational studies are eligible.
* Have known active Central Nervous System (CNS) metastases and / or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they have stable CNS disease for at least 4 weeks prior to enrollment and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking ≤ 10 mg/day of Prednisone or its equivalent. All patients with carcinomatous meningitis are excluded regardless of clinical stability. Current or prior use of immunosuppressive medication within 28 days prior to IMP treatment start, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids as mentioned above.
* Major surgical procedure within 28 days prior to IMP treatment start.
* Have ongoing AEs not recovered to grade 1 or better due to a previously administered agent.

(Note: If patients received major surgery, they must have recovered adequately from the toxicity and / or complications from the intervention prior to starting therapy.)

* Preexisting peripheral sensory neuropathy (> grade 1).
* Uncontrolled diabetes mellitus.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:
* Patients with vitiligo or alopecia
* Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Patients without active disease in the last 5 years prior to IMP treatment start may be included but only after consultation with the sponsor
* Patients with celiac disease controlled by diet alone
* Patients with an HIV detectable viral load at known history of HIV-1 or 2.
* Have active Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV). In patients with a history of HBV or HCV, patients with detectable viral loads will be excluded.
* Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
* Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
* History of allogeneic organ transplant.
* Receipt of live attenuated vaccine (active influenza vaccines excluded) within 30 days prior to IMP treatment start. Note: Patients, if enrolled, should not receive live vaccine during trial treatment and up to 30 days after the last IMP dose.
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness / social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Met any of the following criteria for cardiac disease:

  * Myocardial infarction or unstable angina pectoris within 6 months of IMP treatment start.
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
  * New York Heart Association (NYHA) class III or greater congestive heart failure or LVEF of < 40%.
* Have active serious infection requiring antibiotics.
* Any medical condition that, in the investigator's or sponsor's opinion, poses an undue risk to the patient's participation in the study.
* Any concurrent drug contraindicated for blocking the effect of Magrolimab; this includes systemic corticosteroids (exceptions see above), Methotrexate, Azathioprine, and Tumor Necrosis Factor (TNF)-α blockers.
* Any concurrent drug contraindicated for use with Cisplatin or Gemcitabine according to the locally approved product information.
* Known hypersensitivity to Magrolimab, Cisplatin, or Gemcitabine, its metabolites, or formulation excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity in Run-in Phase | End of cycle 1 (day 21)
  Incidence of DLTs in participants of the safety run-in phase
Proportion of participants with any AEs of severity grade 3 or higher | Up to 6 months after IMP dose initiation
  Proportion of participants with any AEs of severity grade 3 or higher according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 over 6 months after IMP dose initiation

SECONDARY OUTCOMES:
Progression-Free Survival | 48 months
  PFS from date of dose initiation as determined by investigator assessment per RECIST, Version 1.1
Duration Of Response | 48 months
  DOR, defined as time from first documentation of complete response or partial response to the earliest date of documented disease progression, per RECIST, Version 1.1, or death from any cause, whichever occurs first, as determined by investigator assessment
Date of dose initiation to death | 48 months
  DOS, defined as date of dose initiation to death from any cause.
Proportion of complete or partial response (ORR) | 48 months
  The proportion of patients who achieve a complete response or partial response (ORR), as measured by response evaluation criteria in solid tumors (RECIST version 1.1, as determined by investigator assessment

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 48 months
  Incidence of AEs including any laboratory abnormalities according to CTCAE, version 5.0
Reported AEs | From start of treatment with IMP until 28 days after the last IMP dose or the initiation of subsequent anticancer therapy, whichever is sooner
  All AEs from start of treatment with IMP until 28 days after the last IMP dose or the initiation of subsequent anticancer therapy, whichever is sooner

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Kiss, Professor, Principal Investigator — Universtary Hospital Insel Bern

IPD SHARING:
Plan to Share IPD: No